CLINICAL TRIAL: NCT03618160
Title: A Double-blind, Placebo-controlled, Randomized, Single Ascending Dose and Multiple Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics Following Subcutaneous Injections of JNJ-64565111 in Healthy Male Japanese Subjects and An Open-label, Single Dose Study to Assess Pharmacokinetics Following Subcutaneous Injections of JNJ-64565111 in Healthy Male Caucasian Subjects
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of Subcutaneous (SC) Injections of JNJ-64565111 in Healthy Male Japanese Participants and to Assess Pharmacokinetics Following Subcutaneous Injections of JNJ-64565111 in Healthy Male Caucasian Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The results of leading Phase 2 trials did not meet all desired endpoints
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108497; 64565111NAS1001 (Other: Janssen Pharmaceutical K.K)
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: SAD (Cohort 1 to 3) (Experimental): Participants in Cohorts 1 to 3 will receive a single Subcutaneous (SC) low, medium, and high dose of JNJ-64565111 or a JNJ-64565111 matched placebo respectively on Day 1, under fasted conditions in healthy Japanese male participants. Doses in subsequent cohorts will be escalated based on review of Principal Investigator and the Sponsor's decision after safety, tolerability review to determine safe and maximum well tolerated dose.
  Interventions: Drug: JNJ-64565111; Drug: Placebo
- Part 2: MAD (Cohort 4 to 6) (Experimental): Participants in Cohorts 4 to 5 will receive weekly multiple SC low and high dose of JNJ-64565111 or a JNJ-64565111 matched placebo respectively on Day 1, under fasted conditions in healthy Japanese male participants. If multiple high dose is judged as not tolerable, additional optional Cohort 6 will be added to Part 2 to investigate the safety, tolerability and PK after administration of multiple medium dose of JNJ-64565111 in healthy Japanese male participants. Doses in subsequent cohorts will be escalated based on review of Principal Investigator and the Sponsor's decision after safety and tolerability review to determine safe and maximum well tolerated dose.
  Interventions: Drug: JNJ-64565111; Drug: Placebo
- Part 3: Single Dose (Cohort 7) (Experimental): Participants in Cohort 7 will receive a single SC medium dose of JNJ-64565111 which may be started (as early as) in parallel with Cohort 3 in Part 1 on Day 1, under fasted conditions in healthy Caucasian male participants. Based on the results from Cohort 1 to 3 in Part 1, the dose of Cohort 7 may be reduced to low dose or increased to high dose.
  Interventions: Drug: JNJ-64565111

INTERVENTIONS:
Drug: JNJ-64565111 — Participants in Cohorts 1 to 3 will receive a single SC low, medium, and high dose of JNJ-64565111 respectively on Day 1, participants in Cohorts 4 to 6 will receive weekly multiple SC low, high and medium dose of JNJ-64565111 respectively on Days 1, 8, 15, and 22, under fasted conditions. Participants in Cohort 7 will receive a single SC medium dose of JNJ-64565111 on Day 1, under fasted conditions.
Drug: Placebo — Participants will receive SC injection of matching placebo on Day 1 in all cohorts of Part 1 and on Days 1, 8, 15, and 22 in Part 2 under fasted conditions.
  Arms: Part 1: SAD (Cohort 1 to 3); Part 2: MAD (Cohort 4 to 6)

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics (PK) of JNJ-64565111 following single and multiple subcutaneous (SC) doses in healthy Japanese male participants.

ELIGIBILITY:
Inclusion Criteria:

* For Part 1 and Part 2, participant must be a Japanese male 20 to 65 years of age, inclusive, at the time of informed consent for screening. For Part 3, participant must be a Caucasian male (defined as white and all of his parents and grandparents are white as determined by participant's verbal report) 20 to 65 years of age, inclusive, at the time of informed consent for screening
* Participant must agree to use an adequate contraception method as deemed appropriate by the investigator; to always use a condom during sexual intercourse (even in case of prior vasectomy), or to remain abstinent, and not to donate sperm during the study and for 90 days after study drug administration. Participants should encourage their female partner to use an effective method of contraception (example, prescription oral contraceptives, contraceptive injections, intrauterine device, or contraceptive patch) in addition to the condom used by the male study participant
* Participant must have a body mass index (BMI) ranging from 25 to 40 kilogram per meter square (kg/m^2), weighing 120 kilogram (kg) or less
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12 lead electrocardiogram (ECG) performed at screening
* Participant must be a non smoker for at least 1 month prior to screening. A positive urine smoking test (cotinine) at screening and/or admission (Day 2) will lead to exclusion

Exclusion Criteria:

* Participant having a history of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiovascular disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), significant pulmonary disease, including bronchospastic respiratory disease, hepatic or renal insufficiency, type 1 diabetes mellitus, type 2 diabetes mellitus (T2DM), diabetic ketoacidosis (DKA), pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study result
* Participant has taken any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, from 14 days before the first dose of the study drug is scheduled until completion of the study
* Participant has received an experimental drug (including investigational vaccines) or used an experimental medical device within 3 months or within a period less than 5 times the drug's half life, whichever is longer, prior to screening
* Participant test positive for human immunodeficiency virus (HIV [positive serology for HIV antigen/antibody]), tests positive for hepatitis B virus surface antigen, or has antibodies to hepatitis C virus (HCV) at screening
* Participant has had major surgery (example, requiring general anesthesia) within 4 months before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study or within 6 months after study drug administration

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The main reason to enroll male participants in this study is to decrease operational difficulties at site level as there is no specific reason to enroll female participants.
Enrollment: 42 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Part 1 and Part 3: Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to Day 35
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product.
Part 1: Maximum Observed Serum Concentration (Cmax) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  Cmax is defined as the maximum observed serum concentration.
Part 1: Actual Sampling Time to Reach Maximum Observed Serum Concentration (Tmax) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  Tmax is defined as the actual sampling time to reach maximum observed serum concentration of JNJ-64565111.
Part 1: Area Under Serum Concentration Curve From Time 0 to Time of the Last Measurable Concentration (AUC[0-Last]) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  AUC(0-Last) is defined as the AUC from time 0 to the time of the last measurable (non-below quantification limit [non-BQL]) serum concentration.
Part 1: Area Under the Serum Concentration-Time Curve From Time 0 to Infinity (AUC[0-Infinity]) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  AUC (0-infinity) is defined as the area under the serum concentration-time curve from time zero to infinite time calculated as the sum of AUC(0-last) and Clast/ lambda (z); wherein AUC(0-last) is area under the serum concentration time curve from time zero to last measurable serum concentration, Clast is the last observed measurable (non-BQL) serum concentration, and lambda (z) is the apparent terminal elimination rate constant.
Part 1: Apparent Terminal Elimination Half-Life (t1/2) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  t1/2 is defined as the apparent terminal elimination half life, and is calculated as 0.693/lambda (z).
Part 1: Apparent Volume of Distribution (V/F) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  V/F is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution after subcutaneous dose (V/F) is influenced by the fraction absorbed and calculated as dose/(lambda (z)*AUC[0-infinity]).
Part 1: Total Apparent Clearance (CL/F) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  CL/F is defined as the total apparent clearance of drug after extravascular administration calculated as: dose divided by AUC[0-infinity].
Part 2: Number of Participants With AEs as a Measure of Safety and Tolerability | Up to Day 72
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product.
Part 2: Maximum Observed Serum Concentration (Cmax) of JNJ-64565111 | Day 1: Predose, 8, 24, 48, 72, 120 hours postdose; Day 22: Predose, 72, 96, 144, 168, 312, 480, 720, 1200 hours postdose
  Cmax is defined as the maximum observed serum concentration.
Part 2: Actual Sampling Time to Reach Maximum Observed Serum Concentration (Tmax) of JNJ-64565111 | Day 1: Predose, 8, 24, 48, 72, 120 hours postdose; Day 22: Predose, 72, 96, 144, 168, 312, 480, 720, 1200 hours postdose
  Tmax is defined as the actual sampling time to reach maximum observed serum concentration of JNJ-64565111.
Part 2: Apparent Terminal Elimination Half-Life (t1/2) of JNJ-64565111 | Day 22: Predose, 72, 96, 144, 168, 312, 480, 720, 1200 hours postdose
  t1/2 is defined as the apparent terminal elimination half life, and is calculated as 0.693/lambda (z).
Part 2: Apparent Volume of Distribution (V/F) of JNJ-64565111 | Day 22: Predose, 72, 96, 144, 168, 312, 480, 720, 1200 hours postdose
  V/F is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution after subcutaneous dose (V/F) is influenced by the fraction absorbed and calculated as dose/(lambda (z)*AUCtau).
Part 2: Total Apparent Clearance (CL/F) of JNJ-64565111 | Day 22: Predose, 72, 96, 144, 168, 312, 480, 720, 1200 hours postdose
  CL/F is the total apparent clearance of drug after extravascular administration calculated as: dose divided by AUCtau.
Part 2: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of JNJ-64565111 | Day 1: Predose, 8, 24, 48, 72, 120, 168 hours postdose; Day 22: 72, 96, 144, 168 hours postdose
  AUCtau is defined as the measure of the serum drug concentration from time zero to end of dosing interval.
Part 2: Observed Serum Concentration Just Prior to the Beginning or the End of a Dosing Interval (Ctrough) of JNJ-64565111 | Day 8: Predose ; Day 15: Predose; Day 22: Predose, 168 hours postdose
  Ctrough is defined as the observed serum concentration just prior to the beginning or the end of a dosing interval.
Part 2: Average Concentration Over the Dosing Interval Tau (T) at Steady State (Caverage,ss) of JNJ-64565111 | Day 22: Predose, 72, 96, 144, 168 hours postdose
  Caverage,ss is defined as area under the serum concentration time curve observed during a dosing interval (tau) at steady state) will be calculated as AUCtau/Tau.
Part 2: Observed Accumulation Index (AR-AUC) of JNJ-64565111 | Day 1: Predose, 8, 24, 48, 72, 120, 168 hours postdose; Day 22: Predose, 72, 96, 144, 168, 312, 480, 720, 1200 hours postdose
  AR-AUC is determined after multiple dose administration of JNJ-64565111 and calculated by using the equation: AUCtau, Day 22 divided by AUCtau, Day 1.

SECONDARY OUTCOMES:
Part 1 and 3: Number of Participants With Anti-Drug Antibodies (ADAs) to JNJ-64565111 | Predose, 144 and 816 hours postdose
  Number of participants with anti-drug antibodies (ADAs) to JNJ-64565111 will be reported.
Part 1 and Part 3: Change From Baseline in Body Weight | Baseline to Day 35
  Change from baseline in body weight will be reported.
Part 1 and Part 3: Change from Baseline in Fasting Plasma Glucose (FPG) Levels | Baseline to Day 35
  Change from baseline in FPG levels will be reported.
Part 1 and Part 3: Change From Baseline in Total Cholesterol | Baseline to Day 35
  Change from baseline in total cholesterol will be reported.
Part 1 and Part 3: Change From Baseline in Low Density Lipoprotein- Cholesterol (LDL-C) | Baseline to Day 35
  Change from baseline in LDL-C will be reported.
Part 1 and Part 3: Change From Baseline in High-Density Lipoprotein-Cholesterol (HDL-C) | Baseline to Day 35
  Change from baseline in HDL-C will be reported.
Part 1 and Part 3: Change From Baseline in Very Low Density Lipoprotein-Cholesterol (VLDL-C) | Baseline to Day 35
  Change from baseline in VLDL-C will be reported.
Part 1 and Part 3: Change From Baseline in Triglycerides | Baseline to Day 35
  Change from baseline in Triglycerides will be reported.
Part 1 and Part 3: Change From Baseline in Free Fatty Acids | Baseline to Day 35
  Change from baseline in free fatty acids will be reported.
Part 2: Number of Participants With Anti-Drug Antibodies (ADAs) to JNJ-64565111 | Predose on Day 1, 8, 15, 22 and then at 144, 480, 720, 1200 hours postdose
  Number of participants with ADAs to JNJ-64565111 will be reported.
Part 2: Change From Baseline in Body Weight | Baseline to Day 72
  Change from baseline in body weight will be reported.
Part 2: Change From Baseline in Fasting Plasma Glucose (FPG) Levels | Baseline to Day 72
  Change from baseline in FPG levels will be reported.
Part 2: Change From Baseline in Total Cholesterol | Baseline to Day 72
  Change from baseline in total cholesterol will be reported.
Part 2: Change From Baseline in Low Density Lipoprotein- Cholesterol (LDL-C) | Baseline to Day 72
  Change from baseline in LDL-C will be reported.
Part 2: Change From Baseline in High-Density Lipoprotein-Choelsterol (HDL-C) | Baseline to Day 72
  Change from baseline in HDL-C will be reported.
Part 2: Change From Baseline in Very Low Density Lipoprotein-Cholesterol (VLDL-C) | Baseline to Day 72
  Change from baseline in VLDL-C will be reported.
Part 2: Change From Baseline in Triglycerides | Baseline to Day 72
  Change from baseline in triglycerides will be reported.
Part 2: Change From Baseline in Free Fatty Acids | Baseline to Day 72
  Change from baseline in free fatty acids will be reported.
Part 3: Maximum Observed Serum Concentration (Cmax) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  Cmax is defined as the maximum observed serum concentration.
Part 3: Actual Sampling Time to Reach Maximum Observed Serum Concentration (Tmax) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  Tmax is defined as the actual sampling time to reach maximum observed serum concentration of JNJ-64565111.
Part 3: Area Under Serum Concentration Curve From Time 0 to Time of the Last Measurable Concentration (AUC[0-Last]) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  AUC(0-Last) is defined as the AUC from time 0 to the time of the last measurable non-below quantification limit serum concentration.
Part 3: Area Under the Serum Concentration-Time Curve From Time 0 to Infinity (AUC[0-Infinity]) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  AUC (0-infinity) is defined as the area under the serum concentration-time curve from time zero to infinite time calculated as the sum of AUC(0-last) and Clast/ lambda (z); wherein AUC(0-last) is area under the serum concentration time curve from time zero to last measurable serum concentration, Clast is the last observed measurable (non-BQL) serum concentration, and lambda (z) is the apparent terminal elimination rate constant.
Part 3: Apparent Terminal Elimination Rate Constant (Lambda [z]) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  Lambda (z) is the apparent terminal elimination rate-constant, estimated by linear regression using the terminal log linear phase of the log transformed concentration vs time curve.
Part 3:Apparent Terminal Elimination Half-Life (t1/2) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  t1/2 is defined the apparent terminal elimination half life, and is calculated as 0.693/lambda (z).
Part 3: Apparent Volume of Distribution (V/F) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  V/F is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution after subcutaneous dose (V/F) is influenced by the fraction absorbed and calculated as dose/(lambda (z)*AUC[0-infinity]).
Part 3: Total Apparent Clearance (CL/F) of JNJ-64565111 | Predose, 1, 2, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 816 hours postdose
  CL/F is defined as the total apparent clearance of drug after extravascular administration calculated as: dose divided by AUC[0-infinity].

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (2):
- Japan (2):
  - Souseikai Hakata Clinic, Fukuoka
  - Sumida Hospital, Tokyo